CLINICAL TRIAL: NCT05919810
Title: The Effects of Oral Probiotics and Herbal Supplementation on the Gut Microbiome and Sebum Excretion Rate in Non-Cystic Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Codex Labs (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CB_Acne_Supp
Record Dates: First submitted 2023-06-16; First posted 2023-06-26 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-05

CONDITIONS: Acne Vulgaris; Acneiform Eruptions; Skin Diseases; Sebaceous Gland Diseases
Keywords: microbiome; probiotics; dietary supplementation
MeSH Terms: conditions — Acne Vulgaris; Acneiform Eruptions; Skin Diseases; Sebaceous Gland Diseases | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic (Experimental): Daily consumption of probiotic
  Interventions: Other: Probiotic
- Oral herbal supplement (Experimental): Daily consumption of oral herbal supplement powder
  Interventions: Dietary Supplement: Oral herbal powder supplement

INTERVENTIONS:
Other: Probiotic — Oral probiotic
  Arms: Probiotic
Dietary Supplement: Oral herbal powder supplement — oral herbal powder
  Arms: Oral herbal supplement

SUMMARY:
The purpose of this study is to evaluates how probiotics and dietary supplementation with an herbal powder can shift the gut microbiome in those with non-cystic acne vulgaris.

DETAILED DESCRIPTION:
The investigators hope to evaluate the effects of oral supplements in changing intestinal health and the gut bacteria in patients with non-cystic acne vulgaris.

Acne is a chronic inflammatory condition that is estimated to affect greater than 85% of the population at some point. While antibiotics are typically used for systemic therapy, it can increase the risk for drug-resistant bacteria and shift the gut microbiome in a negative way. On the other hand, probiotics and dietary supplementation have been shown to support the gut microbiome.

In this study, participants will be randomized to either receiving a probiotic or powder supplement.

This means that participants will have an equal chance of receiving either product as half of the participants will be randomized to receive only oral probiotic, and the other half will receive oral supplement powder.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 12 years of age until 45 years of age
* The presence of mild to moderate acne based on investigator global assessment.
* Presence of at least 10 inflammatory lesions and at least 5 non-inflammatory lesions

Exclusion Criteria:

* The presence of severe acne as noted by the investigator global assessment.
* Those who are unwilling to discontinue oral probiotic-based supplementation, or supplement ingredients found in the study's oral product 1 month prior to enrollment.
* Those who are unwilling to discontinue topical antibiotics and topical benzoyl peroxide for 2 weeks prior to enrollment
* Those who are unwilling to keep their facial regimen the same throughout the study
* Individuals who have been on an oral antibiotic for acne within the previous one month.
* Individuals who are pregnant or breastfeeding.
* Individuals who have changed any of their hormonal based contraception or therapies within 3 months prior to joining the study.
* Individuals on oral contraceptive pills or progesterone or estrogen containing therapies
* Use of isotretinoin within the three months prior to enrollment.
* Individuals on finasteride or dutasteride
* Current tobacco smoker or a tobacco smoking history

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Gut microbiome composition of short chain fatty acid producing bacteria | 8 weeks
  Change on the relative abundance of Akkermansia mucinaphila and Facelibacterium pruasntizii
Stool acetate levels | 8 weeks
  Assess the short chain fatty acid stool acetate levels

SECONDARY OUTCOMES:
Change in salivary progesterone levels | 4 weeks
  Progesterone and 17-OH progesterone levels
Change in salivary progesterone levels | 8 weeks
  Progesterone and 17-OH progesterone levels

OTHER OUTCOMES:
Total lesion count | 4 weeks
  Safety endpoint to count inflammatory and non-inflammatory lesions
Total lesion count | 8 weeks
  Safety endpoint to count inflammatory and non-inflammatory lesions

CONTACTS AND LOCATIONS:
Overall Officials: Raja Sivamani, MD MS AP, Principal Investigator — Principal Investigator
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Min M, Afzal N, Maloh J, Dulai AS, Ahmad N, Pinzauti D, Sivamani RK. Prospective Comparative Study of an Oral Synbiotic and a Myoinositol-Based Herbal Supplement in Modifying Hormone Levels and the Gut Microbiome in Non-cystic Acne. Dermatol Ther (Heidelb). 2025 Jun;15(6):1331-1350. doi: 10.1007/s13555-025-01411-4. Epub 2025 Apr 18. PMID 40246799